CLINICAL TRIAL: NCT00002233
Title: A Phase II, 48-Week, Uncontrolled, Open-Label Study Designed to Evaluate the Safety and Efficacy of Quadruple Antiretroviral Therapy (EPIVIR, Abacavir, Amprenavir, and Indinavir) in Subjects Acutely Infected With HIV-1
Brief Title: A Study of a Combination of Four Drugs in Patients With Recent HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 264K; COLA 2012
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; CD4 Lymphocyte Count; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; abacavir; amprenavir; Lamivudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Lamivudine

SUMMARY:
The purpose of this study is to see if it is safe to give a combination of four anti-HIV drugs to patients recently infected with HIV who have never received anti-HIV treatment. The effects of this combination of drugs on the immune system and the level of HIV in the body are studied also. The four-drug combination includes lamivudine, abacavir, amprenavir, and indinavir.

DETAILED DESCRIPTION:
Patients receive a four-drug regimen consisting of two nucleoside reverse transcriptase inhibitors (3TC and abacavir) and two protease inhibitors (amprenavir and indinavir) for a minimum of 48 weeks. At specified time points, patients undergo physical assessments and efficacy evaluations which include plasma HIV-1 RNA measurements and CD4 cell counts. Depending on the immunologic and virologic status of the patient, further testing may be done to determine whether quadruple drug therapy can attain undetectable viral levels.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed with caution and/or careful monitoring:

* Drugs which may interact at CYP3A4 (e.g., alprazolam, carbamazepine, codeine, clarithromycin, dapsone, diazepam, diltiazem, erythromycin, estrogens, fluvastatin, glucocorticoids, imipramine, lidocaine, lovastatin, nifedipine, phenobarbital, phenytoin, simvastatin, and warfarin).
* Drugs that inhibit cytosolic alcohol dehydrogenase (e.g., ethanol, disulfiram, chlorzoxazone, chlorpromazine, isoniazid, and chloral hydrate).
* Drugs known to affect renal tubular secretion (e.g., probenecid or cimetidine), cause liver toxicity, or induce myelosuppression.

Patients must have:

* Documented and confirmed acute HIV-1 infection.
* No prior exposure to antiretroviral treatment.
* Ability to comply with the investigational nature of the study for a minimum of 48 weeks.
* Consent of parent or guardian if under the age of 18.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* A clinical diagnosis of AIDS, excluding CD4+ cell counts less than 200/mm3.
* A serious medical condition such as diabetes, congestive heart failure, cardiomyopathy, or other cardiac dysfunction that, in the opinion of the investigator, compromises the safety of the patient.
* Institutionalized or mentally disabled.
* Inability to comply with the dosing schedule and protocol evaluations for reasons other than those specified.

Concurrent Medication:

Excluded:

* Concurrent therapy with rifampin, rifabutin, terfenadine, astemizole, ketoconazole, itraconazole, cisapride, triazolam, midazolam, quinidine, amiodarone, and/or ergotamine/dihydroergotamine-containing regimens.
* Foscarnet or therapy with other agents with documented in vitro or in vivo activity against HIV-1.
* Medications known to induce or inhibit hepatic cytochrome P450 enzyme systems.
* Vitamin E supplements.

Concurrent Treatment:

Excluded:

* Dependence on blood transfusions.
* Other investigational treatments.

Patients with the following prior conditions are excluded:

* A history of clinically relevant pancreatitis or hepatitis within 6 months of study entry.
* A history of inflammatory bowel disease or malignancy, intestinal ischemia, malabsorption, or other gastrointestinal dysfunction that might interfere with drug absorption or render the patient unable to take oral medication.
* An unexplained fever above 38.5 Celsius for more than 14 days within 30 days of study entry.
* A history of coagulopathy.

Prior Medication:

Excluded:

* Prior exposure to antiretroviral therapy.
* Therapy with immunomodulating agents such as systemic corticosteroids, interleukins, thalidomide, anti-cytokine agents or interferons, cytotoxic chemotherapeutic agents, or anti-oxidants within 30 days of study entry.

Prior Treatment:

Excluded:

- Radiation therapy within 30 days of study entry.

Risk Behavior:

Excluded:

Alcohol or illicit drug use which, in the opinion of the investigator, may interfere with ability to comply with the dosing schedule and protocol evaluations.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Aaron Diamond AIDS Rsch Ctr / Rockefeller Univ, New York, New York
  - Miriam Hosp / Family Healthcare Ctr at SSTAR, Providence, Rhode Island